CLINICAL TRIAL: NCT00634582
Title: Phase II Trial of Zemplar (19-nor-1 a,25-Dihydroxyvitamin D2, Paricalcitol Capsule) on Bony Remodeling in Advanced Androgen-Insensitive Prostate Cancer
Brief Title: Paricalcitol in Treating Patients With Advanced Prostate Cancer and Bone Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00004564; P30CA012197 (NIH); CCCWFU-85107
Record Dates: First submitted 2008-03-12; First posted 2008-03-13 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Metastatic Cancer; Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer; bone metastases
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — paricalcitol; Immunoenzyme Techniques; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: paricalcitol
Other: immunoenzyme technique
Other: laboratory biomarker analysis
Procedure: dual x-ray absorptometry
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Paricalcitol may help prostate cancer cells become more like normal cells, and to grow and spread more slowly. It may also stop the growth of tumor cells in bone.

PURPOSE: This phase II trial is studying how well paricalcitol works in treating patients with advanced prostate cancer and bone metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To explore the relationship between paricalcitol therapy and markers of bone formation in patients with androgen-refractory, advanced prostate cancer with bone metastases.

Secondary

* To explore the relationship between paricalcitol therapy and markers of bone resorption in these patients.

OUTLINE: Patients receive oral paricalcitol once daily for 10 weeks in the absence of unacceptable toxicity.

Patients undergo blood sample collection periodically to determine markers of bone formation and resorption by ELISA; parathyroid hormone (PTH) levels by immunometric assay; prostate-specific antigen (PSA) levels by immunoassay; and 25-hydroxyvitamin D and 1,25(OH)_2D levels by radioimmunoassay.

Patients also undergo a bone densitometry (DEXA scan) at baseline and at 10 weeks to assess changes in bone strength.

Quality of life is assessed prior to, during, and after completion of treatment. Questionnaires include the Pain Inventory, the Brief Pain Inventory, the Functional Assessment of Cancer Therapy-G (FACT-G), and the Analgesic Use Diary (Narcotic Pain Medication Logbook).

After completion of study treatment, patients are followed every 6 months for 1 year.

ELIGIBILITY:
Inclusion:

* Histologically or cytologically confirmed advanced adenocarcinoma of the prostate

  - Radiographically proven bone metastasis from prostate cancer
* Androgen refractory disease (including anti-androgen withdrawal)
* Secondary hyperparathyroidism, defined as two parathyroid hormone (PTH) values > 70 pg/mL, 14 days apart
* ECOG performance status 0-2
* Leukocytes ≥ 3,000/μL
* Absolute neutrophil count ≥ 1,500/μL
* Platelets ≥ 100,000/μL
* Total bilirubin normal
* AST/ALT ≤ 2.5 times upper limit of normal
* Creatinine clearance ≥ 60 mL/min
* Calcium normal
* 25-hydroxyvitamin D (25-OHD) ≥ 20 ng/mL
* 1,25(OH)_2D normal
* Patients with serum 25-OHD indicative of vitamin D insufficiency are eligible provided they are treated with ergocalciferol to raise 25-OHD levels to 20 ng/mL prior to paricalcitol therapy
* More than 8 weeks since prior bisphosphonates
* More than 2 weeks since prior palliative radiotherapy
* More than 4 weeks since other prior therapy
* No more than one prior taxane-containing chemotherapy regimen for metastatic disease
* Multiple lines of prior therapy with hormonal agents allowed
* Concurrent corticosteroids allowed provided the dose remains stable during the study period

Exclusion:

* Underlying metabolic bone disease or vitamin D deficiency
* History of hypercalcemia
* Concurrent uncontrolled illness or co-morbid condition (including psychiatric illness) that would interfere with study compliance
* Concurrent ergocalciferol supplementation
* Concurrent chemotherapy or hormonal therapy
* Concurrent investigational or commercial agents for the malignancy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary G. Schwartz, MD, PhD, MPH, Study Chair — Wake Forest University Health Sciences; Mebea Aklilu, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Paricalcitol: Paricalcitol capsules (Zemplar, Abbott) will be given on day 1 at 1 micrograms by mouth and continue daily for 16 weeks if all conditions for continuation are met
Period: Overall Study
Arm/Group | Paricalcitol
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Paricalcitol
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.8 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Markers (i.e., Serum Parathyroid Hormone [PTH], Bone-specific Alkaline Phosphatase, and Osteocalcin) That Are Surrogates for Fracture Risk and Are Associated With Increased Bone Pain, Morbidity, and Mortality From Prostate Cancer
Time Frame: 16 weeks
Population: This trial was closed for slow accrual. For cost reasons, analysis was to be done in a batch size never reached, so the analysis was not done.
Arm/Group | Paricalcitol
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Paricalcitol
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paricalcitol (N=2)
Pain (General disorders) | 1 (1)
hyponatremia (Investigations) | 1 (1)
Edema: limb (Vascular disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Syncope (fainting) (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paricalcitol (N=2)
low Platelets (Investigations) | 1 (1)
Low Hemoglobin (Investigations) | 2 (2)
Anorexia (General disorders) | 1 (1)
Alkaline phosphatase (Investigations) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Neurology (Nervous system disorders) | 1 (2)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
hyperglycemia (Investigations) | 2 (2)
hypocalcemia (Investigations) | 1 (1)
hypoalbuminemia (Investigations) | 1 (1)
serum glutamic pyruvic transaminase (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
serum glutamic oxaloacetic transaminase (Investigations) | 2 (2)
Fever without neutropenia (General disorders) | 1 (1)
Cardiac Arrhythmia - Other (Cardiac disorders) | 1 (1)
Edema: limb (Vascular disorders) | 1 (1)
Confusion (General disorders) | 1 (1)
Ataxia (General disorders) | 1 (1)
Pain: Back (General disorders) | 1 (1)
Pain: Bone (General disorders) | 1 (1)
Flushing (General disorders) | 1 (1)
Voice changes (General disorders) | 1 (1)
Lymphopenia (Investigations) | 1 (1)
Muscle weakness (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes